CLINICAL TRIAL: NCT06815848
Title: Venous Drainage of the Craniocervical Junction: a Retrospective Anatomical Study
Brief Title: Venous Drainage of the Craniocervical Junction: a Retrospective Anatomical Study (SVCR MR1)
Acronym: SVCR MR1
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0312 - SVCR MR1
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-12

CONDITIONS: Study of Venous Drainage of the Cranio-Cervical Junction Using MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to examine the feasibility of distinctly visualizing the different cervical venous networks (subcutaneous, muscular, extra-canalicular, and intra-canalicular) using dedicated magnetic resonance imaging (MRI) sequences. Theoretically, these venous networks contribute to the complex distribution of blood drainage in the cervical region, but their precise identification on imaging remains challenging.The objectives of this research are twofold: first, to assess the ability of MRI to differentiate each venous network, thereby enhancing the anatomical and functional understanding of this region; and second, to explore the possibility of grouping patients according to the predominant venous network, which could reveal significant physiological variations and specific anatomical profiles.The results could not only refine the diagnosis of cervical vascular pathologies but also guide targeted therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated with a social security system
* Age >18 years
* Patient who underwent a T1 Angio-MRI with gradient echo and contrast agent of the cranio-cervical region, regardless of the indication, at the Brest University Hospital between 01/01/2019 and 01/11/2024

Exclusion Criteria:

* Patients under judicial protection (guardianship, curatorship, etc.) Refusal to participate (expressed opposition) History of venous occlusive pathology OR vascular pathology such as cerebral or spinal AVM/FAV History of posterior cranial fossa surgery OR surgical approach to the posterior cervical spine History of radiotherapy/chemotherapy/any known vein-toxic therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Brest University Hospital who underwent a cranio-cervical MRI with injected T1 GRE sequence between January 1, 2019, and November 1, 2024.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of venous vessel in the four venous networks (subcutaneous, muscular, extra-canal, and intra-canal). | at the time of inclusion
  Determine, for each patient, which cervical venous network is dominant and identify whether each patient exhibits all four venous networks (subcutaneous, muscular, extra-canal, and intra-canal).

SECONDARY OUTCOMES:
Number of vessel in each groups | at the time of inclusion
  Assess the relative significance of each identified venous network.
number of vessel on the left and the right in one patient | at the time of inclusion
  Examine whether there is a dominance of venous drainage on the right or left side in the same patient

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement